CLINICAL TRIAL: NCT03271658
Title: Development of an Individualized, Web-Based Life Support Decision Aid (eLSDA) Concerning Goals of Care for the Seriously Ill Patient
Brief Title: Mixed Methods Study Web-based Life Support Decision Aid
Acronym: eLSDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatchewan Health Research Foundation (Other)
Responsible Party: Principal Investigator, Anh Pham, Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: BEH12334
Record Dates: First submitted 2017-08-29; First posted 2017-09-05 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Clinical Decision-Making
Keywords: patient decision aid; end-of-life care; shared decision making; informed decision; decision-making; clinical decision-making; web-based decision aid; palliative; critical care; nursing

STUDY DESIGN:
Intervention Model Description: This study includes 1) a randomized controlled trial and 2) an embedded observational qualitative study. The randomized control trial will compare a convenience cohort of participants who receive usual care (approximately n=60 patients or patient/surrogate pairs) to a cohort of participants who receive the intervention (approximately n=60 patients or patient/surrogate pairs).
Who Masked: Participant, Care Provider
Masking Description: The doctor will not be told which intervention was used with the patient. The patient/family are told that they will have one of two ways to see the information about life support, but are blind to which is classified as the study intervention and standard care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patient/family are randomized to either the active intervention (web based life support patient decision aid - eLSDA and decision coaching) or usual care comparison.
  Interventions: Behavioral: Web based life support patient decision aid; Behavioral: Decision coaching
- Usual Care Comparison (No Intervention): Patients may also randomized to review current web based resources provided by the health region for seriously ill patients.

INTERVENTIONS:
Behavioral: Web based life support patient decision aid — The web-based life support decision aid (eLSDA) was adapted from a print-based decision aid. The eLSDA includes information on the pros and cons of both life support and comfort care. The eLSDA lays out the decision about life support for an individual patient/family in a logical stepwise fashion to permit discussion, ask questions, and permit reflection on each step. At the end of the eLSDA, unmet decision-making needs are identified to seek support from the healthcare team.
  Other Names: eLSDA
  Arms: Intervention
Behavioral: Decision coaching — During the interactive process of using the eLSDA, the study nurse provides decision coaching for patient/family, specifically a facilitated values clarification exercise.
  Other Names: expert facilitation
  Arms: Intervention

SUMMARY:
Patients and families want to be involved in healthcare decisions. When the decision-making process does not engage older patients and their families, the care provided does not match patient preferences or meet their needs. Healthcare teams can collaborate to support patients and families facing difficult healthcare decisions, such as decisions about the use of technology used to keep a person alive when they are critically ill. Tools called patient decision aids are used in many health care settings to help patients and families understand their options and figure out the benefits and harms of a treatment to decide what is right for them. The healthcare team can make sure that patients understand the information provided, give them opportunities to ask questions, and help them talk more about the decision with others. This research study is trialing a web based patient decision aid class of intervention. It is anticipated that 120 hospitalized, seriously ill, older adult patients/ families and their healthcare professionals will be recruited. The study will determine if the intervention can improve dialogue about whether life sustaining technology for seriously ill older patients. The findings will contribute to what is already known about overcoming challenges to involving patients and families with a goal of keeping patients and families at the centre of decisions about their health.

DETAILED DESCRIPTION:
A concurrent mixed method study of a life support decision aid (eLSDA) intends to prepare hospitalized, seriously ill older adult patients and their families to participate in shared decision-making. The study includes 1) randomized controlled trial and 2) a qualitative (naturalistic observation) study. The experimental study compares a convenience cohort of participants who receive usual care (n=60 patients or patient/surrogate pairs) to a cohort of participants who receive the intervention (n=60 patients or patient/surrogate pairs). The investigators intend to measure a) knowledge of life-sustaining technologies, b) clarity of values, c) congruence between documented physician's orders and patient choice, d) decisional conflict, and e) quality of communication. For the intervention group only, investigators will measure comprehensibility and acceptability of the eLSDA. The observational qualitative study derived from naturalistic observation will involve participant observation to examine dialogue about life support between hospitalized, seriously ill older adult patients, families and their healthcare professionals. Quantitative and qualitative data will be collected to better understand the comprehensibility, acceptability, usability, feasibility and impact of the eLSDA used in routine clinical practice.

Questionnaires, patient/family/physician discussions and web based tool viewing will be completed in a hospital setting. The investigator will administer pre-intervention questionnaires to the participants, which will take approximately 15 minutes. Participants will then be randomized to groups, and be invited to use the web based eLSDA or usual care materials on a laptop computer or tablet (30 minutes). This will be followed by post-intervention questionnaires in a second interview (15 minutes). Physicians and nurses/social workers will be asked to complete a survey to examine the barriers to discussions about goals of care (15 minutes). The investigator will also fill out the chart abstraction tool after the participants give consent.

ELIGIBILITY:
Inclusion Criteria:

* Potential users of eLSDA, which are those who are hospitalized, seriously ill, older patients, their families, and their health care providers.
* Age 55 + with one or more of the following diseases:

  1. Chronic obstructive lung disease
  2. Congestive heart failure
  3. Cirrhosis
  4. Cancer
  5. End-stage dementia
  6. Renal failure
* Any patient 70 + admitted to the hospital from the community because of an acute medical or surgical condition.
* Any patient 55 - 69 years of age admitted to the hospital, who has high likelihood of death in the next 6 months, in the opinion of the treating physician.

Exclusion Criteria:

* People who are not hospitalized or do not have family members that are hospitalized and are not a potential user of the eLSDA.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2017-01-29 (Actual); Study Completion 2017-01-29 (Actual)

PRIMARY OUTCOMES:
Acceptability & Usability of the eLSDA | up to 15 minutes
  The acceptability and usability is assessed by conducting an Acceptability Survey which asks participants 8 validated questions about the use, amount of information, length, clarity, balance in presentation, willingness to recommend to others and overall suitability for decision making. The intervention will be considered acceptable if score of the acceptability survey exceeds 80%.

SECONDARY OUTCOMES:
Knowledge about life-sustaining technologies | up to 15 minutes
  This knowledge of life-sustaining technologies will be measured after using the eLSDA using the self-report questionnaire. The knowledge questionnaire was developed for this study based on the eLSDA to test users' knowledge of life-sustaining technologies.
Clarity of values regarding life-sustaining technologies | up to 30 minutes
  The patient's values will be collected in the eLSDA.
Congruence between the documented physician's orders and patient choice | up to 5 minutes
  Congruence between documented physician orders and patient choice when participants use the eLSDA and/or based on patient communication during the discussion with their physician will be reported as simple agreement: (Yes/No)
Feasibility of Evaluation Process | up to 30 minutes
  The measures of feasibility are established by the rate of completion of the eLSDA, debriefing and study procedures. The study will be considered feasible if 60% of those approached agreed to participate in the study; >75% of participants discuss the decision about life support during the encounter, <5% of the participants are distressed by the eLSDA, and 80% of participants complete data collection.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Kryworuchko, PhD RN CNCC, Principal Investigator — University of British Columbia; Wanda Martin, PhD RN, Study Director — University of Saskatchewan; Donna Goodridge, Study Chair — University of Saskatchewan; Petrina McGrath, Study Chair — Saskatoon Health Region; Karen Levesque, Study Chair — Saskatoon Health Region
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] The Change Foundation. Consumers and Canadian Health Care Trending Analysis 2004. The Change Foundation: Toronto. 2005.
- [Background] Heyland DK, Groll D, Rocker G, Dodek P, Gafni A, Tranmer J, Pichora D, Lazar N, Kutsogiannis J, Shortt S, Lam M; Canadian Researchers at the End of Life Network (CARENET). End-of-life care in acute care hospitals in Canada: a quality finish? J Palliat Care. 2005 Autumn;21(3):142-50. PMID 16334968
- [Background] Elwyn G, O'Connor A, Stacey D, Volk R, Edwards A, Coulter A, Thomson R, Barratt A, Barry M, Bernstein S, Butow P, Clarke A, Entwistle V, Feldman-Stewart D, Holmes-Rovner M, Llewellyn-Thomas H, Moumjid N, Mulley A, Ruland C, Sepucha K, Sykes A, Whelan T; International Patient Decision Aids Standards (IPDAS) Collaboration. Developing a quality criteria framework for patient decision aids: online international Delphi consensus process. BMJ. 2006 Aug 26;333(7565):417. doi: 10.1136/bmj.38926.629329.AE. Epub 2006 Aug 14. PMID 16908462
- [Background] O'Connor AM, Graham ID, Visser A. Implementing shared decision making in diverse health care systems: the role of patient decision aids. Patient Educ Couns. 2005 Jun;57(3):247-9. doi: 10.1016/j.pec.2005.04.010. No abstract available. PMID 15893205
- See also: Decide Together Survey - Life Support Decision Aid — https://fluidsurveys.usask.ca/s/decidetogether/